CLINICAL TRIAL: NCT04173793
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of AK102 in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study of PCSK9 Inhibitor AK102 in Patients With Heterozygous Familial Hypercholesterolemia (HeFH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: AD Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK102-201
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: HeFH; LDL-C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AK102 450 mg (Experimental): Participants received AK102 450 mg subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- AK102 300 mg (Experimental): Participants received AK102 300 mg subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- AK102 150 mg (Experimental): Participants received AK102 150 mg subcutaneous injection once every 2 weeks (Q2W) for 12 weeks
  Interventions: Drug: AK102; Drug: Statins and/or Ezetimibe
- Placebo Q4W (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: Placebo; Drug: Statins and/or Ezetimibe
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks
  Interventions: Drug: Placebo; Drug: Statins and/or Ezetimibe

INTERVENTIONS:
Drug: AK102 — Administered by subcutaneous injection
  Arms: AK102 150 mg; AK102 300 mg; AK102 450 mg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo Q4W
Drug: Statins and/or Ezetimibe — Lipid-lowering therapies

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multicenter study to evaluate the safety and efficacy of AK102 in patients with heterozygous familial hypercholesterolemia (HeFH).The primary objective of this study is to evaluate the efficacy of AK102 in patients with HeFH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with heterozygous familial hypercholesterolemia diagnosed by genetic confirmation or clinical diagnosis criteria.
* Stable on pre-existing, lipid-lowering therapies (statins with or without ezetimibe) for at least 4 weeks with no planned medication or dose change for the duration of study participation.
* Fasting Low-Density Lipoprotein Cholesterol (LDL-C) ≥ 70 mg/dL in patients with history of Atherosclerotic Cardiovascular Disease (ASCVD) or Fasting Low-Density Lipoprotein Cholesterol (LDL-C) ≥ 100 mg/dL in patients without history of Atherosclerotic Cardiovascular Disease (ASCVD).
* Fasting triglycerides ≤ 400 mg/dL.
* Body weight ≥ 40kg.

Key Exclusion Criteria:

* Subjects with homozygous FH (clinically or by genotyping).
* Receipt of LDL apheresis within 12 months prior to the first dose of Investigational product.
* Receipt of Lomitapide or Mipomersen within 5 months prior to the first dose of Investigational product.
* Prior use of PCSK9 inhibitors.
* Creatine kinase (CK) >3 times of the upper limit of normal (ULN).
* Aspartate Aminotransferase (AST) ≥ 2 x ULN.
* Estimated Glomerular Filtration Rate (eGFR)≤ 30 mL/min/1.73m^2.
* Thyroid-Stimulating Hormone (TSH)> 1.5 x ULN or <1 x LLN.
* Type 1 diabetes, or type 2 diabetes that is or poorly controlled（HbA1c> 8.5%).
* Subjects with untreated or active chronic hepatitis B or active hepatitis C virus infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 12 | At baseline and week 12

SECONDARY OUTCOMES:
Percent change from baseline in low-density lipoprotein cholesterol (LDL-C) | From baseline through 12 weeks
Percent change from baseline in high-density lipoprotein cholesterol (HDL-C) | From baseline through 12 weeks
Percent change from baseline in non High-density lipoprotein (non-HDL) cholesterol | From baseline through 12 weeks
Percent change from baseline in serum Triglyceride (TG) cholesterol | From baseline through 12 weeks
Percent change from baseline in Apolipoprotein B (Apo B) | From baseline through 12 weeks
Percent change from baseline in Apolipoprotein A-I (ApoA-I) | From baseline through 12 weeks
Percent change from baseline in Lipoprotein(a) [Lp-(a)] | From baseline through 12 weeks
Percent change from baseline in Total Cholesterol(TC) | From baseline through 12 weeks
Incidence of treatment-emergent adverse events | From baseline through 12 weeks
Serum concentrations of AK102 | From baseline through 12 weeks
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline through 12 weeks
  The immunogenicity of AK102 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies.
Change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Principal Investigator — Peking Union Medical College Hospital; Yujie Zhou, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No